CLINICAL TRIAL: NCT05387473
Title: Towards PREcision MEdicine for Osteoarthritis: Added Value of Cognitive Behavioural Therapy for Insomnia.
Brief Title: Added Value of Cognitive Behavioural Therapy for Insomnia in Persons With Knee Osteoarthritis
Acronym: PREMEO
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: KU Leuven (Other); Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Jo Nijs, Professor, Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FWO TBM T000521N
Record Dates: First submitted 2022-05-12; First posted 2022-05-24 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Knee; Insomnia
Keywords: sleep initiation and maintenance problems; Arthritis; Pain; Sleep Disorders, Intrinsic; Dyssomnias; Sleep Wake Disorder
MeSH Terms: conditions — Osteoarthritis, Knee; Sleep Initiation and Maintenance Disorders; Arthritis; Pain; Sleep Disorders, Intrinsic; Dyssomnias; Sleep Wake Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cognitive behavioral therapy for insomnia (CBT-I) integrated in best-evidence usual care (CBTi-UC) (Experimental): 18 individual sessions provided by physiotherapists, over 14 weeks.
  Interventions: Behavioral: Cognitive behavioral therapy for insomnia (CBT-I) integrated in best-evidence usual care (CBTi-UC)
- Best-evidence usual care (UC) plus information sessions (Active Comparator): 18 individual sessions provided by physiotherapists, over 14 weeks.
  Interventions: Behavioral: Best-evidence usual care (UC) plus information sessions

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy for insomnia (CBT-I) integrated in best-evidence usual care (CBTi-UC) — In the first two weeks, the participants will receive three sessions of education and advice based on current best-practice guidelines. In the following three weeks, the participants will be provided with once weekly exercise therapy and once weekly CBT-I. This is then spread out more over the next five weeks in which participants will receive once weekly sessions of either CBT-I or exercise therapy in alternating order. In the last four weeks of the intervention period, the participants will receive once weekly exercise therapy.
  Arms: cognitive behavioral therapy for insomnia (CBT-I) integrated in best-evidence usual care (CBTi-UC)
Behavioral: Best-evidence usual care (UC) plus information sessions — In the first two weeks, the participants will receive three sessions of education and advice based on current best-practice guidelines. In the following three weeks, the participants will be provided with once weekly exercise therapy and once weekly general information sessions (general education sessions in line with recommendations from best-practice guidelines and recent evidence). This is then spread out more over the next five weeks in which participants will receive once weekly sessions of either CBT-I or exercise therapy in alternating order. In the last four weeks of the intervention period, the participants will receive once weekly exercise therapy.
  Arms: Best-evidence usual care (UC) plus information sessions

SUMMARY:
Knee osteoarthritis (KOA) is the leading and fastest increasing cause of disability in older adults. It is a serious health issue related with a high health care utilisation. The first-line KOA management is nonsurgical care, with education and exercise therapy as key elements. Nevertheless, treatment effects of exercise therapy and behavioral pain management on improvements in pain, function and quality of life are small to moderate at best. This shows that there is an urgent need for better KOA care. The innovative solution may lie in thinking beyond joints, by targeting KOA subgroups through comorbidity-specific interventions, which fits well in the global move towards precision medicine. With a prevalence rate up to 50%, the presence of insomnia symptoms is a highly prevalent KOA comorbidity, contributing to symptom severity. If left untreated, it represents a barrier for effective conservative management. Since insomnia is nowadays hardly addressed in the often joint-targeted KOA care, the scientific objectives of the study are to assess 1) if cognitive behavioral therapy for insomnia (CBT-I) integrated in best-evidence usual care, consisting of education and exercise therapy, (CBTi-UC) is more effective than best-evidence usual care alone (UC), i.e. education and exercise therapy, at 6 months follow-up in improving clinical outcomes and 2) if CBTi-UC is more cost-effective than UC in KOA patients with comorbid insomnia.

ELIGIBILITY:
Inclusion Criteria:

45 years old or older

Being a fluent Dutch speaker

Commits to study requirements

Knee Osteoarthritis classified using the American college of Rheumatology criteria (Knee pain + 3/6 for diagnosis):

* age>50
* morning stiffness <30 minutes
* crepitus
* bony tenderness
* bony enlargement
* no palpable warmth

Insomnia diagnosis using the DSM-5 criteria:

* No shiftwork
* No severe untreated sleep disorders
* For at least >3 days / week for >3 months: >30 minutes sleep latency and/or >30 minutes awake after sleep onset and/or early-morning awakening with inability to return to sleep AND associated daytime symptoms

Knee pain nominated by the patient as 3 or higher on a visual analogue scale on most days of the last 3 months

Informed consent

Exclusion Criteria:

Treatment with supervised exercise therapy or joint infiltrations (e.g., corticosteroids, hyaluronic acid) or CBT-I in the preceding six months

Change in any psychiatric or psychological treatment the last 3m or planned during the study period

Concurrent intense psychological treatment (weekly basis)

BMI >30

Mini-Mental state examination score of 23 or lower

Being on the waiting list for a knee replacement or having received knee replacement on symptomatic side

Any contra-indication for exercise therapy

Existing diagnose that has impact on sleep and patients are therefore unlikely to respond to CBT-I: any rheumatological condition (e.g. rheumatoid arthritis, Lupus, Sjogren's syndrome); any neurological conditions (e.g. stroke, Multiple sclerosis, Parkinson's disease), dementia or receiving cholinesterase inhibitors; cancer diagnosis in the past year and receiving chemotherapy or radiation therapy in the past year; Long-COVID or inpatient treatment for congestive heart failure within the prior six months.

Having severe underlying sleep disorder (obstructive sleep apnea over AHI >15, periodic leg movement disorder, restless leg syndrome, sleep-wake cycle disturbance, rapid eye movement behavior disorder)

Being pregnant or given birth in the preceding year

Having an external/ physical factor that limits the opportunity to sleep (E.g. newborn)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in Pain subscale Knee injury and Osteoarthritis Outcome Score | 6 months after the end of therapy
  The pain subscale of the Knee injury and Osteoarthritis Outcome Score (KOOS) will be used as primary outcome to assess change in pain. The KOOS shows adequate content validity, internal consistency, reliability, content validity and responsiveness for age and condition relevant subscales.
  The pain scale consists of 9 items. A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems). The total score ranges from 0 to 36.

SECONDARY OUTCOMES:
Change in Pain subscale Knee injury and Osteoarthritis Outcome Score | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, and 12 months after the end of therapy
  The pain subscale of the Knee injury and Osteoarthritis Outcome Score (KOOS) will be used as primary outcome to assess change in pain. The KOOS shows adequate content validity, internal consistency, reliability, content validity and responsiveness for age and condition relevant subscales.
  The pain scale consists of 9 items. A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems). The total score ranges from 0 to 36.
Change in impact of pain on functioning | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  The Brief Pain Inventory (BPI) evaluates the impact of pain on functioning. The BPI measures how much pain interferes with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others, and sleep on an 11-point Numeric Rating Scale (ranging from 0-10).
Change in self-reported central sensitization symptoms | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  The Central Sensitization Inventory investigates self-reported central sensitization symptoms. Score ranges from 0 to 100, with higher scores indicating more self-reported symptoms of central sensitization.
Change in sleep quality | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  The Pittsburg Sleep Quality Index investigates self-reported perceived sleep quality. Score ranges from 0 to 21, 0 indicating no difficulty and 21 indicating severe sleep difficulties.
Change in Dysfunctional Beliefs and Attitudes about Sleep | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  The Dysfunctional Beliefs and Attitudes about Sleep questionnaire investigates self-reported dysfunctional beliefs and attitudes about sleep. Score ranges from 0 to 10. Scores above 4 indicate unrealistic expectations for sleep or unrealistic thoughts about sleep.
Change in sleep propensity | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  The Epworth Sleepiness Scale investigates self-reported sleep propensity. Score ranges from 0 to 24, with 0 indicating normal daytime sleepiness and 24 indicating severe excessive daytime sleepiness.
Change in pain-related fear of movement | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  The Tampa Scale for Kinesiophobia - 17 item version investigates pain-related fear of movement and (re)injury. Each item is scored on a 4-point Likert Scale, ranging from one ("strongly disagree") to four ("strongly agree"). The total score ranges between 17 and 68, with higher values reflecting greater fear of movement
Change in physical function | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  Change in physical function is assessed with the function in daily living subscale of the Knee injury. and Osteoarthritis Outcome Score
Global assessment | After 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  The patient global assessment is a recommended question in clinical trials of rehabilitation interventions for OA and it measures the improvement or deterioration of their condition since baseline, and therefore since the intervention has started. It will be assessed by patients on a 7-point Likert scale (very much improved, much improved, slightly improved, not changed, slightly worsened, much worsened, and vastly worsened).
Change in physical activity and sleep behaviour | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  Using Fitbit Sense, physical activity measures such as the number of steps as well as sleep parameters will be retrieved with custom-made algorithms to quantify daily movement/sleep behaviours
Change in physical activity and sleep behaviour during intervention | after intervention week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12, week 13, week 14
  Using Fitbit Sense, physical activity measures such as the number of steps as well as sleep parameters will be retrieved with custom-made algorithms to quantify daily movement/sleep behaviours
Change in pain intensity | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  The Numeric Rating Scale for pain assesses the intensity of pain. It is an 11-point scale that requires the patient to select a number ranging from zero ("no pain") to ten ("worst possible pain"). The average and worst pain intensity in last week is questioned.
Change in pain intensity during intervention | Bafter intervention week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12, week 13, week 14
  The Numeric Rating Scale for pain assesses the intensity of pain. It is an 11-point scale that requires the patient to select a number ranging from zero ("no pain") to ten ("worst possible pain"). The average and worst pain intensity in last week is questioned.
Change in insomnia Severity | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  The Insomnia Severity Index investigates self-reported insomnia severity. Score ranges from 0 to 28, with 0 indicating no clinically significant insomnia and 28 indicating severe clinical insomnia.
Change in insomnia Severity during intervention | after intervention week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12, week 13, week 14
  The Insomnia Severity Index investigates self-reported insomnia severity. Score ranges from 0 to 28, with 0 indicating no clinically significant insomnia and 28 indicating severe clinical insomnia.
Change in fatigue severity | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  The Brugmann Fatigue Scale investigates self-reported fatigue severity. Score ranges from 0 to 24, with higher scores indicating higher subjective levels of fatigue.
Change in fatigue severity during intervention | after intervention week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12, week 13, week 14
  The Brugmann Fatigue Scale investigates self-reported fatigue severity. Score ranges from 0 to 24, with higher scores indicating higher subjective levels of fatigue.
Change in pain catastrophizing | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapy and 12 months after the end of therapy
  The Pain Catastrophizing Scale assesses negative thoughts and feelings when experiencing pain. Each item is scored from zero ("not at all") to four ("all the time"). Its total score ranges between 0 and 52, with a higher total score indicating higher levels of pain catastrophizing.
Change in pain catastrophizing during intervention | after intervention week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12, week 13, week 14
  The Pain Catastrophizing Scale assesses negative thoughts and feelings when experiencing pain. Each item is scored from zero ("not at all") to four ("all the time"). Its total score ranges between 0 and 52, with a higher total score indicating higher levels of pain catastrophizing.
Change in anxiety and Depression | Baseline, after 14 weeks (post-intervention), 3 months after the end of therapy, 6 months after the end of therapyand 12 months after the end of therapy
  The Hospital Anxiety and Depression rating scale investigates self-reported affective symptoms. Score ranges from 0 to 21, with 0 indicating absence of depression or anxiety and 21 indicating the presence of depression or anxiety.
Change in anxiety and depression during intervention | after intervention week 1, week 2, week 3, week 4, week 5, week 6, week 7, week 8, week 9, week 10, week 11, week 12, week 13, week 14
  The Hospital Anxiety and Depression rating scale investigates self-reported affective symptoms. Score ranges from 0 to 21, with 0 indicating absence of depression or anxiety and 21 indicating the presence of depression or anxiety.
Change in Pressure Pain Thresholds | Baseline, after 14 weeks (post-intervention), and 12 months after the end of therapy
  Pressure Pain Thresholds are measured with a digital pressure algometer (Wagner Instruments), both at symptomatic level (knee) and at remote sites (i.e. secondary hyperalgesia).
Change in objective sleep assessed with polysomnography (PSG) | Baseline, after 14 weeks (post-intervention)
  Participants will be monitored in the comfort of their own home by ambulatory PSG, one night at echt timepoint. PSG will provide sleep related outcomes (time in bed, total sleep time, sleep onset latency, wake duration after sleep onset, early morning awakening, sleep staging N1, N2, N3, REM in durations and % of total sleep time, sleep efficiency, respiratory parameters, myoclonic activity).
Change in biomarkers for inflammation by blood analysis | Baseline, after 14 weeks (post-intervention), and 12 months after the end of therapy
  A relevant panel of biomarkers for chronic low-grade inflammation, modulation of inflammation and pain will be investigated (ultra-sensitivity ELISA for hsCRP, interleukin (IL)1β, IL1RA, IL6, IL8, IL10, MCP1, tumor necrosis factor (TNF-α, sTNFR1&2, CXCL-10, CX3CL1). Blood sampling will be performed at the hospital after overnight fasting.
Change in physical performance | Baseline, after 14 weeks (post-intervention), and 12 months after the end of therapy
  30sec chair stand test to test leg strength and endurance.While monitoring the participant's performance to ensure proper form, the tester silently counts the completion of each correct stand. The score is the total number of stands within 30 seconds
Change in health care use | Baseline, after 14 weeks (post-intervention), and 12 months after the end of therapy
  Health care use (including co-interventions) will be recorded using the Medical Consumption Questionnaire, a generic instrument for measuring total, (in-)direct medical consumption. This questionnaire is easy-to-use and generates valid data.
Change in productivity cost | Baseline, after 14 weeks (post-intervention), and 12 months after the end of therapy
  The Productivity Cost Questionnaire will be used to obtain data regarding productivity losses. This questionnaire is easy-to-use and generate valid data.
Change in health-related quality of life | Baseline, after 14 weeks (post-intervention), and 12 months after the end of therapy
  The EQ-5D-5L will be used to assess health-related quality of life and to calculated utility health states for the cost-utility analysis. The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS).
  The descriptive system comprises five dimensions, with each dimension consisting of 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. Higher scores indicate a higher quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Jo Nijs, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Department Rehabilitation Science, Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No